CLINICAL TRIAL: NCT04178551
Title: Consortium to Disseminate and Understand Implementation of Opioid Use Disorder Treatment (PII 19-321)
Brief Title: Consortium to Disseminate and Understand Implementation of Opioid Use Disorder Treatment
Acronym: CONDUIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIX 19-001
Record Dates: First submitted 2019-11-21; First posted 2019-11-26 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Opioid Medication Assisted Treatment
Keywords: Opioid Medication Assisted Treatment; Addiction, Opioid
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: The VHA Consortium to Disseminate and Understand Implementation of Opioid Use Disorder Treatment (CONDUIT) will improve access to evidence-based MOUD and advance the science of implementation by providing an integrated, multidisciplinary approach to implementation of evidence-based MOUD across the continuum of care in VHA. CONDUIT implementation teams incorporate expertise from addiction medicine and addiction psychiatry, primary care and hospital medicine, implementation science and health economics. The foundation of CONDUIT's implementation activities are the structured interactions between external facilitation teams and internal facilitation teams. A core set of internal facilitation activities will be used across all facilitation teams, and external facilitation teams will use additional activities based on the needs of their sites or clinical settings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Implementation Facilitation (Other): The foundation of CONDUIT's implementation activities are the structured interactions between external facilitation teams and internal facilitation teams. A core set of internal facilitation activities will be used across all facilitation teams, and external facilitation teams will use additional activities based on the needs of their sites or clinical settings.
  Interventions: Other: Implementation Facilitation
- Pre-Implementation (Other): The pre-implementation period was a period of needs assessment and information-gathering and served as a within-subject comparison condition.
  Interventions: Other: Implementation Facilitation

INTERVENTIONS:
Other: Implementation Facilitation — The foundation of CONDUIT's implementation activities are the structured interactions between external facilitation teams and internal facilitation teams. A core set of internal facilitation activities will be used across all facilitation teams, and external facilitation teams will use additional activities based on the needs of their sites or clinical settings.
  The pre-implementation period served as a comparison condition
  Other Names: Pre-implementation

SUMMARY:
Opioid use disorder (OUD) is a major cause of illness and death among Veterans for which effective treatment is a major priority of the Veterans Health Administration (VHA). Expanding access to alternatives to opioid medications for chronic pain management is also a leading priority. Effective medications for OUD (MOUD) are available, but their availability and use among Veterans varies across VHA. The aims of this study are to pull together the efforts of six individual pilot projects into a single project. The purpose of combining the projects is to maximize the value of the individual projects to VHA and to provide information to guide strategies to increase access and use of MOUD and alternative therapies for pain in VHA nationally. The researchers leading the individual projects will make use of their partnerships with Veterans Integrated Service Network (VISN) leaders in order to develop a combined effort toward increased dissemination and use of MOUD that spans 9 VISNs and 63 sites.

DETAILED DESCRIPTION:
Opioid use disorder (OUD) is a major cause of morbidity and mortality among Veterans and a high-priority target for quality improvement in the Veterans Health Administration (VHA). Effective medications for OUD (MOUD) are available but uptake of them has been highly variable across VHA. Additionally, VHA has been at the forefront in the U.S. in promoting alternative therapies for pain, but these are not consistently available to Veterans in great need of them: those with chronic pain and harmful opioid use. VHA, through its Office of Mental Health and Suicide Prevention, has made access to MOUD for all Veterans who need it a system-wide priority. However, successful implementation of complex care processes that face myriad barriers requires intentional, structured, evidence-based implementation efforts carried out by expert teams in close partnership with local leadership.

As such, the overarching goal of this project - the Consortium to Disseminate and Understand Implementation of Opioid Use Disorder Treatment (CONDUIT) -- is to unite six inter-related VISN/QUERI pilot Partnered Implementation Initiative projects in a concerted effort to improve access to MOUD among Veterans with OUD and access to alternative therapies for pain in 63 VHA sites spanning nine VISNs. CONDUIT will span four critical care settings in the OUD continuum of care: Primary Care; Specialty Care; Acute Care (inpatient and Emergency Department); and Telehealth. These efforts will be connected by Veteran Engagement, Implementation, and Quantitative/Economic Cores that will help CONDUIT teams harmonize on metrics, processes and outcomes. There will also be a Strategic Advisory Group composed of Operations leaders and Veterans that will help CONDUIT remain maximally aligned with VHA and Veteran priorities. CONDUIT will also offer sites the opportunity to implement new evidence-based practices (i.e. ones that were not part of initial launch) in the latter half of the project period.

The methods deployed by each of the CONDUIT teams will be similar: expert "external facilitation" teams will lead partnered "internal facilitation" teams at local sites in a process called "Implementation Facilitation (IF)" - a multi-component suite of tools aimed to help the sites effectively adopt evidence-based practices. The six projects piloted and systematically modified IF strategies in Phase 1 and now propose to disseminate those sharpened strategies on a national scale over the next three years, including new VISNs and dozens of additional sites. In terms of evaluation, CONDUIT will use well-established formative evaluation methods to assess the effectiveness of and to drive refinements to the IF strategies. Additionally, CONDUIT will use cutting edge quantitative methods to assess the impact the work on important clinical targets and to assess the value of the work in terms of costs vs. benefits. Throughout the project period, teams will develop and refine products such as patient and provider educational materials, prescribing and communication guides, and clinic operations manuals. These evaluation and product development efforts will prime successful scale-up and dissemination efforts throughout VHA.

ELIGIBILITY:
Inclusion Criteria:

-All Veterans on prescribed opioid treatment and/or with opioid use disorder who are enrolled at participating implementation sites.

Exclusion Criteria:

-None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C Becker, MD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (11):
- United States (11):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Boise VA Medical Center, Boise, ID, Boise, Idaho
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa
  - Maine VA Medical Center, Augusta, ME, Augusta, Maine
  - VA Central Western Massachusetts Healthcare System, Leeds, MA, Leeds, Massachusetts
  - Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC, Columbia, South Carolina
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individual projects within CONDUIT conducted outreach to VA sites that might benefit from implementation facilitation strategies to support medications for opioid use disorder. Sites opted in/out to receive implementation facilitation. VA Facility Sites were enrolled in the study; patients and providers were not considered enrolled.
Pre-assignment Details: In this study, the intervention occurred at the site level. Site was the level of analysis. Sites advanced from the pre-implementation to implementation phase upon agreement by internal and external facilitation teams.
Units Other Than Participants: VA Facility Sites
Groups:
- Implementation Facilitation: The foundation of CONDUIT's implementation activities are the structured interactions between external facilitation teams and internal facilitation teams. A core set of internal facilitation activities will be used across all facilitation teams, and external facilitation teams will use additional activities based on the needs of their sites or clinical settings.
  Implementation Facilitation: The foundation of CONDUIT's implementation activities are the structured interactions between external facilitation teams and internal facilitation teams. A core set of internal facilitation activities will be used across all facilitation teams, and external facilitation teams will use additional activities based on the needs of their sites or clinical settings.
Period: Pre-Implementation (12 Months)
Arm/Group | Implementation Facilitation
Started | NA; 63 VA Facility Sites (The study was implemented at the site level; therefore individual patients were not characterized. Participants were not assigned to Arm/Groups)
Completed (Number of sites who entered implementation phase following pre-implementation.) | NA; 46 VA Facility Sites (Participants were not assigned to Arm/Groups)
Not Completed | NA; 17 VA Facility Sites
Period: Implementation Facilitation (6-18 Mos)
Arm/Group | Implementation Facilitation
Started | NA; 46 VA Facility Sites (The study was implemented at the site level; therefore individual patients were not characterized. Participants were not assigned to Arm/Groups)
Completed | NA; 46 VA Facility Sites (Participants were not assigned to Arm/Groups)
Not Completed | NA; 0 VA Facility Sites

BASELINE CHARACTERISTICS:
Population: Sites participating in study - this baseline data was not collected
Groups:
- Comparison Cohort: Sites served as their own comparisons.
- Total: Total of all reporting groups
Arm/Group | Implementation Facilitation | Comparison Cohort | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Within Participating Sites With OUD Initiating MOUD During the Implementation Facilitation Period in Implementation Sites. This Will be Compared to Pre-implementation.
Description: Data will be extracted from patients electronic health records and reported at the site level. The denominator for this measure is the number of patients within participating sites eligible to receive MOUD at the site during the target period. This outcome will be compared to pre-implementation.
Time Frame: The implementation period varies by site and will likely range from 6 months to 18 months. The pre-implementation is the 12-month period before implementation.
Measure: Number; unit: patients within participating sites
Groups:
- Implementation Facilitation Period: Implementation Facilitation: The foundation of CONDUIT's implementation activities are the structured interactions between external facilitation teams and internal facilitation teams. A core set of internal facilitation activities will be used across all facilitation teams, and external facilitation teams will use additional activities based on the needs of their sites or clinical settings.
  The start date of the implementation facilitation period for each site was reported by the study PI.
- Pre-Implementation Period: Pre-implementation period defined as the 12 months prior to the implementation start date for each site.
Arm/Group | Implementation Facilitation Period | Pre-Implementation Period
Number analyzed (Participants) | 5127 | 3261
patients within participating sites | 2116 | 974

2. Primary Outcome: Number of Patients Within Participating Sites With OUD Retained on MOUD at 90 Days During the Implementation Period (i.e. Treatment Retention). This Will be Compared to Pre-implementation.
Description: Data will be extracted from patients electronic health records. The denominator for this measure is the number of patients within participating sites receiving MOUD at the time of the site-specific implementation periods.
Time Frame: as for outcome 1
Population: Among Veterans/patients with MOUD initiation, we assessed continued MOUD use, identified as prescription fills for 90 days with no lapses > 30 days. Patients identified as initiating MOUD treatment in a Substance Use Disorder (SUD) clinic were excluded. Patients are counted as retained if they have at least 90 days between first and last SUD visit within phase, without a break > 30 days.
Measure: Number; unit: patients within participating sites
Groups:
- Implementation Facilitation Period: The foundation of CONDUIT's implementation activities are the structured interactions between external facilitation teams and internal facilitation teams. A core set of internal facilitation activities will be used across all facilitation teams, and external facilitation teams will use additional activities based on the needs of their sites or clinical settings.
  Implementation Facilitation: The foundation of CONDUIT's implementation activities are the structured interactions between external facilitation teams and internal facilitation teams. A core set of internal facilitation activities will be used across all facilitation teams, and external facilitation teams will use additional activities based on the needs of their sites or clinical settings.
Arm/Group | Implementation Facilitation Period | Pre-Implementation Period
Number analyzed (Participants) | 1846 | 727
patients within participating sites | 1017 | 357

3. Primary Outcome: Number of Providers Prescribing MOUD During Implementation
Description: The number of prescribing providers will be determined by electronic health record. This is a frequency count. The outcome will be compared to pre-implementation.
Time Frame: as for outcome 1
Population: Prescribers are considered active and having an X-waiver in phase if they held an x-waiver any time from the first day of the month the phase started to the last day of the month the phase ended and had prescribed buprenorphine any time in the 6 months prior.
  Prescribers are considered having an X-waiver (i.e., eligible to prescribe buprenorphine) in phase if they held an x-waiver any time from the first day of the month the phase started to the last day of the month the phase ended.
Measure: Number; unit: prescribers in participating sites
Arm/Group | Implementation Facilitation Period | Pre-Implementation Period
Number analyzed (Participants) | 1554 | 1128
prescribers in participating sites | 474 | 258

4. Primary Outcome: Number of Unique Implementation Strategies Used as Measured by the Expert Recommendations for Implementing Change (ERIC) Survey
Description: Number of unique implementation strategies.
Time Frame: The survey was administered 3-4 months following the start of the study as a baseline measure for comparison to follow-up.
Population: Respondents to ERIC survey
Measure: Number; unit: Number implementation strategies
Arm/Group | Implementation Facilitation Period
Number analyzed (Participants) | 24
Number implementation strategies | 6

5. Primary Outcome: Number of Providers With X-waiver During the Implementation Period
Description: The outcome will be measured by electronic health records. This is a frequency count of providers with X-waivers (for eligibility to prescribe buprenorphine) during the implementation phase. It will be compared to pre-implementation.
Time Frame: The implementation period varies by site and will likely range from 6 months to 18 months. Pre-implementation is the 12 months prior to implementation.
Population: Prescriber data comes from a custom extract similar to the X-Waiver/buprenorphine prescriber report, which details providers holding a Drug Enforcement Administration (DEA) X-waiver on a monthly level.
Measure: Number; unit: count of prescribers
Arm/Group | Implementation Facilitation Period | Pre-Implementation Period
Number analyzed (Participants) | 1554 | 1128
count of prescribers | 1554 | 1128

6. Primary Outcome: Count of Implementation Strategies as Measured by the Expert Recommendations for Implementing Change (ERIC) Survey
Description: Number of unique implementation strategies .
Time Frame: The survey was administered 12 months following a baseline measure (equivalent to 16 months following the start of the CONDUIT trial)
Population: Respondents to ERIC survey
Measure: Number; unit: Number implementation strategies
Arm/Group | Implementation Facilitation Period
Number analyzed (Participants) | 41
Number implementation strategies | 10

7. Secondary Outcome: Percentage of Patients With OUD Who Experienced a Fatal Opioid-related or Other Drug Overdose During Implementation
Description: Data will be extracted from patients electronic health records. Patients experienced an overdose if we observe any recorded overdose events within the first 12 months of the phase. Overdoses are not exclusively opioid-related, but include only fatal events. Counts in the first 12 months of the implementation facilitation period are compared to counts in the 12-month pre-implementation period.
Time Frame: This outcome is measured for first 12 months of the implementation phase and compared to the measure for the pre-implementation period.
Population: We used the suicide navigator data from PERC to identify fatal and non-fatal overdose events. Cohort is defined as veterans who had a visit with an associated OUD diagnosis during the relevant phases. Patients must be observed in phase for at least 30 days. Overdose - Veterans experienced an overdose if we find any recorded overdose events within the first 12 months of the phase. Overdoses are not exclusively opioid-related, and include only fatal events.
Measure: Count of Participants; unit: Participants
Arm/Group | Implementation Facilitation Period | Pre-Implementation Period
Number analyzed (Participants) | 6289 | 5325
Participants | 5 | 6

8. Secondary Outcome: Percentage of Patients With OUD Who Experienced Opioid-related or Other Drug Overdose During Implementation
Description: Data will be extracted from patients electronic health records. Patients experienced an overdose if we observe any recorded overdose events within the first 12 months of the phase. Overdoses are not exclusively opioid-related, and include both fatal and nonfatal events. Counts in the first 12 months of the implementation facilitation period are compared to counts in the 12-month pre-implementation period.
Time Frame: This outcome is measured for first 12 months of the implementation phase and is compared to the 12-month pre-implementation period.
Population: We used the suicide navigator data from PERC to identify fatal and non-fatal overdose events. Cohort is defined as veterans who had a visit with an associated OUD diagnosis during the relevant phases. Patients must be observed in phase for at least 30 days. Overdose - Veterans experienced an overdose if we find any recorded overdose events within the first 12 months of the phase. Overdoses are not exclusively opioid-related, and include both fatal and non-fatal events.
Measure: Count of Participants; unit: Participants
Arm/Group | Implementation Facilitation Period | Pre-Implementation Period
Number analyzed (Participants) | 6289 | 5325
Participants | 272 | 188

9. Secondary Outcome: Use of Sedative Prescriptions During Implementation Among Patients With OUD
Description: This is the count/percentage of people exposed to any sedative prescriptions as determined by patients' electronic health records.
Time Frame: The implementation period varies by site and will likely range from 6 months to 18 months. This outcome is compared to 12-month the pre-implementation period.
Population: Patients were counted as having a prescription for benzodiazepines if they were dispensed at least 1 prescription of benzodiazepines at any time during the phase. Patients were included in the numerator if they had a qualifying prescription during the phase. They were included in the denominator for each phase in which they had a qualifying opioid use disorder diagnosis.
Measure: Count of Participants; unit: Participants
Arm/Group | Implementation Facilitation Period | Pre-Implementation Period
Number analyzed (Participants) | 4872 | 3037
Participants | 1538 | 888

ADVERSE EVENTS:
Time Frame: The intervention for this quality improvement (QI) study was conducted at the site level. Implementation facilitation strategies promoted usual care. Adverse events were not tracked.
Description: This study did not involve an experimental intervention, nor direct intervention with patients. Therefore we did not track adverse events at the patient level.
Groups:
- Comparison Cohort: All other sites in VA not receiving CONDUIT implementation support or participating in other dedicated MOUD implementation activities during the same time period
Arm/Group | Implementation Facilitation | Comparison Cohort
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT04178551/Prot_SAP_000.pdf